CLINICAL TRIAL: NCT06588257
Title: Acceptability of the Human Papillomavirus (HPV) Vaccine and Anal HPV in Transgender Women (TGW) and Men Who Have Sex With Men (MSM): A Pilot Study
Brief Title: Acceptability of the HPV Vaccine and Anal HPV in Transgender Women and Men Who Have Sex With Men: A Pilot Study
Acronym: HPVac
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, FLORENCIA MARINA CAHN, MD, Fundación Huésped
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FH-79
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HPV
Keywords: HPV; MSM; TGW; Acceptability; vaccine

STUDY DESIGN:
Intervention Model Description: A pilot study of mixed quantitative and qualitative methodology is proposed. A prospective cohort of 100 men who have sex with men and transgender women, with and without HIV will be organized at Fundación Huésped to study acceptability of HPV vaccine and effect of HPV vaccine on anal HPV infection. Moreover, 20 people from the cohort along with 5 additional people who shall not agree to receive the HPV vaccine will participate in in depth interviews. (qualitative component).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Men who have sex with men with HIV (Other): Evaluate the acceptability, uptake, and completion of HPV vaccination.
  Interventions: Biological: Non-infectious adjuvanted recombinant nonavalent HPV vaccine
- Transgender women with HIV (Other): Evaluate the acceptability, uptake, and completion of HPV vaccination.
  Interventions: Biological: Non-infectious adjuvanted recombinant nonavalent HPV vaccine
- Men who have sex with men without HIV (Other): Evaluate the acceptability, uptake, and completion of HPV vaccination.
  Interventions: Biological: Non-infectious adjuvanted recombinant nonavalent HPV vaccine
- Transgender women without HIV (Other): Evaluate the acceptability, uptake, and completion of HPV vaccination.
  Interventions: Biological: Non-infectious adjuvanted recombinant nonavalent HPV vaccine

INTERVENTIONS:
Biological: Non-infectious adjuvanted recombinant nonavalent HPV vaccine — Non-infectious adjuvanted recombinant nonavalent HPV vaccine. Three doses (0, 2, 6 months). (Trade name GARDASIL 9 -MSD).

SUMMARY:
Protocol Title: "Acceptability of the Human Papillomavirus (HPV) Vaccine and Anal HPV in Transgender Women (TGW) and Men Who Have Sex with Men (MSM): A Pilot Study.

DETAILED DESCRIPTION:
Protocol Number: FH-79

Study Objetives:

* Evaluate the acceptability, uptake, and completion of HPV vaccination.
* Determine the baseline prevalence (before HPV vaccination) and incidence of vaccine-specific genotypes of nonavalent HPV in the anus (anatomical site) after vaccination.
* Determine the initial prevalence (before HPV vaccination) and incidence of anal cytological lesions after HPV vaccination.-
* Determine the initial prevalence (before HPV vaccination) and incidence of oral and anogenital lesions associated with HPV, according to physical examination, after HPV vaccination.
* Analyze barriers and facilitators to the acceptability, uptake, and completion of HPV vaccination from the perspective of MSM and TGW.

Patient Population: MSM (men who have sex with men) and TGW (transgender woman)

Study design: Phase IV. Longitudinal and prospective study for which a cohort of 100 MSM (men who have sex with men)and TGW (transgender woman) will be formed at Fundación Huésped. Pilot study of mixed quantitative and qualitative methodology.

Regimens: Non-infectious adjuvanted recombinant nonavalent HPV vaccine. Three doses (0, 2, 6 months). (Trade name GARDASIL 9 -MSD), Duration: 12 months

Sample size: 105 subjects

ELIGIBILITY:
Inclusion Criteria:

* Accept participation in the study by signing informed consent
* Age ≥18 years old
* People who consider themselves men who have sex with men or transgender women
* All eligible people with HIV must meet the following:

  1. stable antiretroviral treatment during the last 6 months and with undetectable viral load (depending on the method used for measurement) within the same period (the participant can bring a laboratory report carried out in the last 6 months). Regarding ART, a change associated with toxicity or simplification may be allowed before 12 weeks of the selection visit, with undetectable VL between 12 weeks and the selection visit; and
  2. CD4 cell count ≥ 200 cells/ml in the last 6 months (participant can bring a laboratory report from the last 6 months)

Exclusion Criteria:

* Have a history or current suspicion of cancer
* Have a known history or current suspicion of high-grade lesion or anal intraepithelial neoplasia related to HPV.
* Have received any dose of HPV vaccine at some time in your life.
* Have received any vaccine in the last 30 days.
* Have a known allergy to any of the components of the HPV vaccine.
* Have a history of a previous severe allergic reaction, regardless of the cause.
* Presenting an acute illness that could alter the study evaluations or could put the participant at risk, according to the researcher's criteria.
* Present chronic or acute immunosuppression (except HIV).
* Have received antineoplastic and immunomodulatory agents or radiotherapy in the 6 months prior to the study or plan to receive these treatments during the study period.
* Having chronic diseases without adequate control.
* Have a diagnosis of ongoing malignant disease.
* Having received immunoglobulins, blood or blood products in the last 3 months.
* Do not participate in another intervention study
* That he is not an employee or first-degree relative of any member of the institution.
* Any condition or clinical situation where it is considered that participation in the study may pose a risk to the patient.* * People with chronic HBV infection, who are receiving treatment and have normal transaminases for the last 6 months can be included in the study. People with chronic HCV infection can enter the study if they have normal transaminases for the last 6 months and do not plan to start treatment during the study. In either case, transaminases can be requested through the study if they are not available.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 101 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of people receiving the first dose of vaccine and of people receiving 3 doses of HPV vaccine among those recruited. | 12 months
  To evaluate uptake HPV vaccination, the proportion of who receiving the first dose of HPV vaccine among those who have entered the study will be estimated, and to assess HPV vaccination completion, the proportion of who receiving three doses of HPV vaccine among those enrolled will be estimated.

SECONDARY OUTCOMES:
Frequency of anal HPV genotypes | 12 months
  To determine the prevalence and incidence of anal HPV genotypes (considering the genotypes in the nonavalent vaccine), HPV genotype from anal samples will be performed to determine the frequency of anal HPV at baseline (day 1), month 6 and month 12.
Frequency of anal HPV related cytologic lesions | 12 months
  To determine the prevalence and incidence of anal HPV-associated cytological lesions, anal cytology will be performed to determine the frequency of anal HPV associated cytological lesions at baseline (day 1), month 6 and month 12.

OTHER OUTCOMES:
Acceptability of HPV vaccine | 12 months
  Through in-depth interviews will evaluate barriers and facilitators, as well as prospective and retrospective acceptability of HPV vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Huésped, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared upon request, 6 months after last patient´s last visit. URL not yet available.